CLINICAL TRIAL: NCT03262909
Title: A Prospective, Open-Label, Multicenter Pivotal Study to Evaluate the Safety and Efficacy of GelrinC® for the Treatment of Symptomatic Articular Cartilage Defects of the Femoral Condyle: A Comparison to Historical Control Microfracture
Brief Title: Pivotal Study to Evaluate the Safety and Efficacy of GelrinC for Treatment of Cartilage Defects
Acronym: SAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Regentis Biomaterials (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-GR-01
Record Dates: First submitted 2017-08-17; First posted 2017-08-25 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Articular Cartilage Defects in the Knee Joint
Keywords: cartilage damage; cartilage defect; chondral lesion; osteochondral lesion; femur; condyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- GelrinC prospective treatment arm (Experimental): Patients will undergo GelrinC implantation.
  Interventions: Device: GelrinC
- Microfracture historical control arm (Other): Microfracture historical control arm
  Interventions: Other: Microfracture historical control arm

INTERVENTIONS:
Device: GelrinC — Patients will undergo GelrinC implantation.
  Arms: GelrinC prospective treatment arm
Other: Microfracture historical control arm — Patients undergo an arthroscopy for evaluation purposes, followed by lesion debridement, and a standard microfracture procedure.
  Arms: Microfracture historical control arm

SUMMARY:
Multicenter, open-label, controlled, non-randomized, double arm trial with a prospective treatment arm (GelrinC). This study compares the efficacy and safety of GelrinC to a historical control arm (microfracture) in the treatment of cartilage defects in the knee.

ELIGIBILITY:
Main Inclusion Criteria:

* Age between 18 and 50.
* Single contained symptomatic lesion located on the femoral condyle of the femur graded as ICRS III or IV with less than 5 mm of bone loss below the subchondral plate.
* Lesion size between 1 and 5 cm2 post debridement, less than or equal to 2.5 cm in diameter.
* BMI ≤35
* Contralateral knee is asymptomatic, stable, fully functional and not medically treated.

Main Exclusion Criteria:

* Presence of an additional grade III or IV symptomatic lesion.
* Recent Osteochondritis Dissecans within 1 year of baseline visit.
* Untreated ACL and/or PCL deficiency or Complex ligamentous instability of the knee.
* Patient is excluded if presenting untreated current meniscal tear or if previous menisci resection was within the last 6 months.
* Previous tendon repair or ligament reconstruction within the last 6 months.
* Failed Mosaicplasty or ACI or MACI or any other cartilage repair product.
* Microfracture performed less than 1 year before baseline visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The change of physical functioning as assessed by patient reported outcome measure (Knee injury and Osteoarthritis Outcome Score (KOOS). | 24 months post-surgery
The change of physical pain as assessed by patient reported outcome measure (Knee injury and Osteoarthritis Outcome Score (KOOS). | 24 months post-surgery

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Horizon Clinical Research, La Mesa, California
  - Hoag Orthopedics, Orange, California
  - University of Colorado, Denver, Colorado
  - Shrock Clinical Research, Fort Lauderdale, Florida
  - Andrews Institute, Gulf Breeze, Florida
  - Jewett Orthopaedic Clinic, Orlando, Florida
  - Optim Orthopedics, Savannah, Georgia
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Peninsula Orthopaedic Associates, Salisbury, Maryland
  - Tria Institute, Bloomington, Minnesota
  - Alpine Orthopedics, Bozeman, Montana
  - University Orthopedics Center, Altoona, Pennsylvania
  - Mansfield Orthopedics, Morrisville, Vermont

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trattnig S, Ohel K, Mlynarik V, Juras V, Zbyn S, Korner A. Morphological and compositional monitoring of a new cell-free cartilage repair hydrogel technology - GelrinC by MR using semi-quantitative MOCART scoring and quantitative T2 index and new zonal T2 index calculation. Osteoarthritis Cartilage. 2015 Dec;23(12):2224-2232. doi: 10.1016/j.joca.2015.07.007. Epub 2015 Jul 14. PMID 26187572
- [Background] Berdichevski A, Shachaf Y, Wechsler R, Seliktar D. Protein composition alters in vivo resorption of PEG-based hydrogels as monitored by contrast-enhanced MRI. Biomaterials. 2015 Feb;42:1-10. doi: 10.1016/j.biomaterials.2014.11.015. Epub 2014 Dec 9. PMID 25542788
- [Derived] Shah SS, Lee S, Mithoefer K. Next-Generation Marrow Stimulation Technology for Cartilage Repair: Basic Science to Clinical Application. JBJS Rev. 2021 Jan 19;9(1):e20.00090. doi: 10.2106/JBJS.RVW.20.00090. PMID 33512974